CLINICAL TRIAL: NCT05008783
Title: A Randomized, Double-blind, Multicenter, Phase III Study Comparing the Efficacy and Safety of AK104 Plus Oxaliplatin and Capecitabine (XELOX) Versus Placebo Plus XELOX as First-line Treatment for Locally Advanced Unresectable or G/GEJ Adenocarcinoma
Brief Title: A Study of AK104 in the First-line Treatment of Locally Advanced Unresectable or Metastatic G/GEJ Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104-302
Record Dates: First submitted 2021-07-30; First posted 2021-08-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AK104 + Oxaliplatin + Capecitabine (Experimental): AK104 in combination with Oxaliplatin and Capecitabine
  Interventions: Drug: AK104
- Placebo + Oxaliplatin + Capecitabine (Placebo Comparator): Placebo in combination with Oxaliplatin and Capecitabine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK104 — AK104 (administered on Day 1 of each cycle, Q3W)+Oxaliplatin (130 mg/m2 intravenous infusion for 2-6 hours on Day 1, Q3W,up to 6 cycles)+ Capecitabine(1000 mg/m2, p.o., Bid, Q3W,up to 6 cycles) . Afterward, AK104 will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W)
  Other Names: Oxaliplatin; Capecitabine
  Arms: AK104 + Oxaliplatin + Capecitabine
Drug: Placebo — Placebo (administered on Day 1 of each cycle, Q3W)+Oxaliplatin (130 mg/m2 intravenous infusion for 2-6 hours on Day 1, Q3W,up to 6 cycles)+ Capecitabine(1000 mg/m2, p.o., Bid, Q3W,up to 6 cycles) . Afterward,Placebo will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W)
  Other Names: Oxaliplatin; Capecitabine
  Arms: Placebo + Oxaliplatin + Capecitabine

SUMMARY:
A randomized, Double-blind, Multicenter, phase III Clinical Study of Comparing the Efficacy and Safety of AK104 Plus Oxaliplatin and Capecitabine (XELOX) Versus Placebo Plus XELOX as First-line Treatment for locally advanced Unresectable or Metastatic Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be enrolled in the study:

  1. Ability to understand and voluntarily sign a written informed consent form (ICF), which must be signed before the specified study procedures required for the study are performed.
  2. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent.
  3. Histopathologically confirmed gastric adenocarcinoma or gastroesophageal junction (GEJ) adenocarcinoma.
  4. Unresectable locally advanced or metastatic gastric adenocarcinoma or GEJ adenocarcinoma.
  5. Subjects have not received prior systemic therapy for locally advanced or metastatic gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction. For subjects who have received prior neoadjuvant/adjuvant chemotherapy or chemoradiotherapy for curative intent, the time between disease progression and last treatment should be at least 6 months.
  6. Subjects have at least one measurable tumor lesion per RECIST v1.1; lesions that received radiotherapy are not selected as target lesions, unless the lesion is the only measurable lesion and has unequivocal progression as judged by imaging, it can be considered as a target lesion.

Exclusion Criteria:

* Subjects who meet any of the following criteria are not eligible to participate in this study:

  1. Subjects with known HER2-positive gastric or GEJ adenocarcinoma.
  2. Histopathology or cytology confirmed other pathological types, such as squamous cell carcinoma, sarcoma, or undifferentiated carcinoma.
  3. Subjects who received palliative local therapy for non-target lesions within 2 weeks prior to the first dose; systemic nonspecific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, etc.) within 2 weeks prior to the first dose; and Chinese herbal medicine or traditional Chinese medicinal products with anti-tumor indications within 2 weeks prior to the first dose.
  4. Subjects who received any prior treatments targeting the mechanism of tumor immunity.
  5. Medical history of gastrointestinal perforation or gastrointestinal fistula within 6 months prior to the first dose. If the perforation or fistula has been treated with resection or repair and the disease has recovered or resolved as judged by the Investigator, enrollment may be allowed.
  6. Active or previously documented inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
  7. Active malignancies within the past 3 years, with the exception of tumors in this study and cured local tumors, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of cervix, carcinoma in situ of breast, localized prostate cancer, etc.
  8. Known active or untreated brain metastases, meningeal metastases, spinal cord compression, or leptomeningeal disease.
  9. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage (≥ 1/month).
  10. Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment, or autoimmune diseases that may relapse or require scheduled treatment as judged by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 610 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (os) | Up to 2 years
  OS in the ITT population.

SECONDARY OUTCOMES:
ORR | Up to 2 years
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1
DCR | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
DoR | Up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
TTR | Up to 2 years
  TTR is defined as the time to response base on RECIST v1.1
PFS | Up to 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first assessed by investigator Per RECIST 1.1
AE | From the subject signs the ICF to 30 days (AE) and 90 days (SAE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.
Observed concentrations of AK104 | From first dose of AK104 through the last dose of AK104, about average of 9 months.
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 30 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (7):
- China (7):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Shen L, Zhang Y, Li Z, Zhang X, Gao X, Liu B, Wang Y, Ba Y, Li N, Zhang R, Zhang J, Chen Y, Chen J, Huang M, Fu Y, Liu M, Liu Z, Zhao J, Li W, Wei J, Li C, Xu N, Guo Z, Cao B, Liu L, Nie P, Wan L, Sheng L, Liu Z, He Y, Gu K, Wu G, Wang W, Zhang F, Qiu W, Guo J, Ying J, Pan H, Xu H, Yuan Y, Bai Y, Wang Z, Xu J, Zhao X, Liu H, Zhang X, Dai W, Xu H, Liu M, Xie L, Tang Y, Jin J, Qu X, Fang X, Huang M, Chen H, Zheng Z, Wang Y, Wang D, Li X, Yu G, Liu H, Zhou Y, Zhong D, Zeng S, Kang M, Wang M, Gao Y, Li W, Wang Z, Zhang M, Zhang J, Li Q, Sun S, Zang A, Lin L, Xie M, Zhuang Z, Zhang T, Yao Z, Lu D, Liu W, Hu M, Wang ZM, Li B, Xia M, Zhang J, Ying X, Pardoll DM, Ji J. First-line cadonilimab plus chemotherapy in HER2-negative advanced gastric or gastroesophageal junction adenocarcinoma: a randomized, double-blind, phase 3 trial. Nat Med. 2025 Apr;31(4):1163-1170. doi: 10.1038/s41591-024-03450-4. Epub 2025 Jan 22. PMID 39843940